CLINICAL TRIAL: NCT03509181
Title: Augmenting Hospitalization for Serious Mental Illness by Targeting Interpretation Bias
Brief Title: Augmenting Hospitalization for Serious Mental Illness: Cognitive Bias Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Courtney Beard, PhD, Assistant Professor, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH113600; R34MH113600 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-26 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Depression; Bipolar Disorder; Anxiety Disorders; Psychiatric Disorder
Keywords: interpretation bias; smartphone; partial hospital
MeSH Terms: conditions — Depression; Bipolar Disorder; Anxiety Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBM (Experimental): Cognitive Bias Modification for Interpretation delivered via smartphone
  Interventions: Behavioral: I-Change; Behavioral: Symptom Tracking
- Symptom Tracking (Active Comparator): Weekly symptom monitoring smartphone app with anxiety and depression symptom scores
  Interventions: Behavioral: Symptom Tracking

INTERVENTIONS:
Behavioral: I-Change — smartphone delivered word-sentence association task that encourages a healthier interpretive style
  Other Names: Cognitive Bias Modification for Interpretation
  Arms: CBM
Behavioral: Symptom Tracking — smartphone delivered self-monitoring of anxiety and depression symptoms

SUMMARY:
Approximately 4.1% of the adult US population meets the criteria for SMI, a mental disorder associated with significant functional impairment. Even when effective, pharmacologic and psychological treatments often leave individuals with SMI with residual symptoms, impairment, and at risk for re-hospitalization and suicide. The month following hospitalization is a particularly risky time; thus, augmentation treatments that can speed up improvement during brief hospital stays, as well as provide a bridge to outpatient care are urgently needed. Thus, the investigators propose to develop an augmentation to psychiatric hospital care (called "I-Change") that can be continued at home following discharge. I-Change targets interpretation bias, the tendency to resolve ambiguous situations negatively. Interpretation bias is a well-established cognitive vulnerability for psychopathology and is associated with poor emotion regulation, rumination, symptom severity, and suicidal ideation. For example, in a psychiatric hospital sample, interpretation bias upon admission accounted for 28% of the variance in treatment response, and predicted suicidal ideation at discharge, controlling for ideation at admission. Although some existing treatments target this mechanism, most notably Cognitive Behavioral Therapy (CBT), they require individuals to be able to recognize their automatic interpretations and use complex techniques to reappraise them. Individuals with SMI who are experiencing symptoms acute enough to require hospitalization are often treatment refractory and may experience particular difficulty applying these techniques. It is therefore critical to more efficiently and effectively engage this target. Over the past 14 years, the Principal Investigator has developed and validated a training task that utilizes repetition and feedback to reinforce a healthier interpretive style. The computer-delivered version of the task was acceptable to an SMI population and led to better treatment response than a placebo task in patients who exhibited interpretation bias at baseline. The investigators seek to develop this task into a personalized smart-phone delivered intervention. The investigators will harness smart-phone technology to enhance skill acquisition and generalization by improving user engagement and prompting participants to complete a session at set times to ensure adequate dosage and spacing of sessions. The investigators will conduct an open trial (n = 16) and a randomized controlled trial (n = 64) to confirm target engagement (improvement in interpretation bias), evaluate the feasibility and acceptability of delivering I-Change during and following discharge from a partial hospital, and examine clinical outcomes (global improvement, functioning) related to changes in interpretation. I-Change is expected to shift interpretation bias, be acceptable to patients with SMI, and lead to greater global improvement compared to a Symptom Tracking control. Results will support a fully-powered effectiveness trial.

DETAILED DESCRIPTION:
Treatment in acute psychiatric hospital settings is brief, and many individuals continue to experience residual symptoms and impairment upon discharge. The months following discharge from hospitalization are particularly risky, as individuals transition from a highly structured and supportive environment to home, acute stressors, and uncertain aftercare. Currently, there are few interventions available to accelerate improvement during brief hospital stays, or to provide a bridge to outpatient care. Thus, there is an urgent need to develop augmentations to hospital care that both more efficiently reduce symptoms during the acute hospital stay and provide continuation of care during the transition to home. Such new interventions are critical to reduce the risk of relapse, re-hospitalization, and suicide in individuals with Serious Mental Illness (SMI).

The long-term goal of this study is to develop effective and scalable interventions that target key mechanisms in psychopathology and are easily implemented in real world settings. The overall objective of this study is to develop a low-intensity augmentation to psychiatric partial hospital care that can be continued during the transition to home. "I-Change", a personalized, smart-phone delivered cognitive bias modification (CBM) treatment, is expected to hasten improvement in pathological cognitive processes and clinical outcomes during hospitalization and following discharge compared to a control. This hypothesis is based on the principal investigator's (PI) 14 years of research developing and testing CBM treatments, including a pilot study of 65 patients attending a partial hospital program that showed excellent feasibility, acceptability, large effects on cognitive bias, and moderate effects on clinical outcomes compared to a placebo control.

I-Change will target the maladaptive interpretative style that maintains emotional disorders. The way in which individuals automatically resolve the countless ambiguous situations encountered each day has a large impact on their affect and behavior. Interpretation bias, the tendency to resolve such ambiguity negatively, is a crucial therapeutic target because it is associated with poor emotion regulation, rumination, symptom severity, suicidal ideation, and treatment response. Although existing treatments target interpretation bias, most notably Cognitive Behavioral Therapy (CBT), they require individuals to recognize their automatic interpretations and use complex techniques to reappraise them. Individuals experiencing symptoms sufficiently acute to require hospital care often experience difficulty applying these techniques. In contrast, the PI validated a computerized training task that utilizes quick, repeated practice and feedback to more efficiently reinforce a healthier interpretive style. Ten studies demonstrate that the task engages interpretation bias and leads to improved clinical outcomes in individuals with mood and anxiety disorders, including a psychiatric hospital sample. The CBM task is highly acceptable and uniquely suited to acute psychiatric settings due to its low complexity and engaging qualities.

Specific Aim 1: Develop a smart-phone delivered intervention to augment hospital care.

This study will harness smart-phone technology to enhance the acquisition of a healthier interpretive style by personalizing the situations presented, prompting participants to complete sessions to ensure adequate dosage, and incorporating features to enhance adherence. Delivery via smart phone increases accessibility of the intervention by overcoming barriers (e.g., transportation, computer access) within the hospital and at home and allows better assessment of outcomes in "real time" via ecological momentary assessment. An Advisory Board of patients, hospital providers, experts in CBM and mobile health technology, and other stakeholders (i.e., directors of acute psychiatric clinics) will inform the development of I-Change.

Specific Aim 2: Obtain pilot data to support a fully-powered randomized controlled trial (RCT), including measures of (a) target engagement (improvement in interpretation bias), (b) feasibility and acceptability of I-Change and procedures for hospital and home delivery, and (c) global improvement and functioning Participants will complete I-Change daily while admitted to the partial hospital and three times per week at home during the 1-month following discharge. Consistent with a precision medicine and RDoC approach, participants will be selected based on baseline level of interpretation bias (not diagnosis). The investigators will first conduct an open trial of I-Change (n = 16) to inform refinements. The investigators will conduct a pilot RCT (n = 64) to obtain data to inform the design of a future trial. Participants will be randomly assigned to I-Change or a Symptom Tracking control and assessed at admission, discharge, 1-month and 3-months following discharge. Obtained data will be compared to a priori benchmarks of feasibility, acceptability, target engagement, and clinical improvement.

The final products of this study will be the I-Change app, RCT protocol, and pilot data to support a future confirmatory effectiveness trial. Achievement of these aims will result in a simple, scalable augmentation to psychiatric partial hospital care that can improve outcomes following hospital care.

ELIGIBILITY:
Inclusion Criteria:

* currently receiving partial hospital care at the study site
* age ≥18
* at least moderate symptom severity (PHQ-9 or GAD-7 score > 10)
* signing a release of information for treatment providers
* a minimal level of interpretation bias (<80% accuracy on the Word Sentence Association Paradigm)

Exclusion Criteria:

* current psychiatric symptoms that would prevent informed consent or understanding of research procedures (e.g., active symptoms of psychosis, mania)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioral Health Partial Hospital/McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will deposit de-identified data in the National Database for Clinical Trials Related to Mental Illness (NDCT) according to NIH guidelines.
Time Frame: every 6 months

REFERENCES:
- [Derived] Beard C, Ramadurai R, McHugh RK, Pollak JP, Bjorgvinsson T. HabitWorks: Development of a CBM-I Smartphone App to Augment and Extend Acute Treatment. Behav Ther. 2021 Mar;52(2):365-378. doi: 10.1016/j.beth.2020.04.013. Epub 2020 Apr 30. PMID 33622506

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Bias Modification + Symptom Tracking: Cognitive Bias Modification for Interpretation delivered via smartphone
  I-Change: smartphone delivered word-sentence association task that encourages a healthier interpretive style
  Symptom Tracking: smartphone delivered self-monitoring of anxiety and depression symptoms
Period: Overall Study
Arm/Group | Cognitive Bias Modification + Symptom Tracking | Symptom Tracking
Started | 34 | 34
Completed | 27 | 31
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Bias Modification + Symptom Tracking | Symptom Tracking | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.29 (10.853) | 32.326 (13.256) | 31.28 (12.064)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant did not identify as Male or Female
  Participants
    number analyzed (Participants) | 33 | 34 | 67
    Female | 21 | 24 | 45
    Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 29 | 57
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Improvement Scale (CGIS)
Description: Self-reported improvement rating. Outcome is number of participants who reported feeling much or very much improved.
Time Frame: Post-treatment (1 month following discharge from hospital) (up to 8 weeks following baseline)
Population: Participants who completed the 1-month follow-up assessment and provided a Clinical Global Improvement rating.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Bias Modification + Symptom Tracking | Symptom Tracking
Number analyzed (Participants) | 25 | 30
Participants | 14 | 20

2. Primary Outcome: 5-item Work and Social Adjustment Scale
Description: The Work and Social Adjustment Scale assesses interference caused by the patient's symptoms in the domains of work, home management, leisure, and family relationships. It includes 5 items each rated from 0 to 8 with total scores ranging from 0 to 40 and higher scores indicating more impairment.
Time Frame: Post-treatment (1 month following discharge from hospital)(up to 8 weeks following baseline)
Population: Participants who completed the 1-month assessment and completed the WSAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Bias Modification + Symptom Tracking | Symptom Tracking
Number analyzed (Participants) | 25 | 30
score on a scale | 19.08 (11.416) | 17.43 (8.617)

3. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) is a 16 item questionnaire that asks about life satisfaction over the past week. Each question is rated on a 5 point scale from 1 (Very Poor) to 5 (Very Good). Scores from the individual items are added together and reported as percentage maximum possible score. The Total Score is reported as percentage maximum possible % Max = Raw-minimum score/maximum score-minimum score. (Raw score minus the minimum possible raw score divided by the maximum possible raw score minus the minimum possible raw score). Higher scores indicate better quality of life.
Time Frame: Post-treatment (1 month following discharge from hospital) (up to 8 weeks following baseline)
Population: Participants who completed the 1-month assessment and the QLESQ (note: missing 1 participant in CBM arm who did not complete the QLESQ).
Measure: Mean (Standard Deviation); unit: percentage of max possible score
Arm/Group | Cognitive Bias Modification + Symptom Tracking | Symptom Tracking
Number analyzed (Participants) | 24 | 30
percentage of max possible score | 45.58 (10.5) | 44.83 (7.40)

ADVERSE EVENTS:
Time Frame: From baseline to 3 months following hospital discharge (up to 4 months).
Arm/Group | Cognitive Bias Modification + Symptom Tracking | Symptom Tracking
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03509181/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03509181/SAP_001.pdf
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03509181/ICF_002.pdf